CLINICAL TRIAL: NCT05401305
Title: Simple Blind, Placebo Controlled, Randomized Safety and Reactogenicity Trial of "Baby-Hib [Vaccine for the Prevention of Infections Caused by Haemophilus Influenzae Type b], Lyophilizate for Preparation of Intramuscular Injection Solution, 0.5 mL/Dose", FSUE SPbSRIVS FMBA of Russia, in Volunteers Aged 18-50
Brief Title: Safety and Reactogenicity Trial of Vaccine for the Prevention of Infections Caused by Haemophilus Influenzae Type b
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Petersburg Research Institute of Vaccines and Sera (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HIB-I-07/19
Record Dates: First submitted 2022-05-27; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Haemophilus Influenzae Infection; Vaccines
Keywords: Haemophilus Influenzae; Haeophilus influenza type b; Vaccine; Hib vaccines; Hib; SPbSRIVS
MeSH Terms: conditions — Haemophilus Infections | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hib vaccine (Experimental): Volunteers will be vaccinated with Vaccine for the prevention of infections caused by Haemophilus influenza type b once intramuscularly at a dose of 0.5 mL.
  Stage I: 5 volunteers Stage II: 25 volunteers
  Interventions: Biological: Vaccine for the prevention of infections caused by Haemophilus influenza type b
- Placebo (Placebo Comparator): Volunteers will receive a placebo once intramuscularly at a dose of 0.5 mL. Stage I: 5 volunteers Stage II: 25 volunteers
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Vaccine for the prevention of infections caused by Haemophilus influenza type b — The vaccine is administered into the region of the deltoid muscle
  Arms: Hib vaccine
Biological: Placebo — The placebo is administered into the region of the deltoid muscle
  Arms: Placebo

SUMMARY:
Trial purpose is to evaluate the safety, tolerability and reactogenicity of the Vaccine for the prevention of infections caused by Haemophilus Influenzae Type b in volunteers aged 18-50.

DETAILED DESCRIPTION:
The trial includes 2 stages (Stage I and Stage II). The aim of the Stage I is to assess the tolerability, reactogenicity and safety of the Hib vaccine in the first 10 volunteers during the first 7 days after vaccination.

The aim of the Stage I is to assess the tolerability, reactogenicity and safety of the Hib vaccine during 28 days after vaccination and also to conduct a comparative assessment of the safety and reactogenicity of the Hib vaccine and placebo during 28 days after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men and women) aged 18-50 years;
* Written informed consent of volunteers to participate in the clinical trial;
* Volunteers not previously vaccinated with any vaccine to prevent infections caused by Haemophilus influenza type b;
* Volunteers able to fulfill requirements of the Protocol (i.e. fill out the patient's diary, come to follow-up visits);
* For fertile women, a negative pregnancy test and consent to observe adequate methods of contraception (if hormonal contraceptives are used, they must be canceled at least 2 months before the start of the trial). All women with childbearing potential must have a negative pregnancy test result during the Data Collection Period. In the course of the trial women should use contraception methods with a reliability exceeding 90 %, or be sterile, or be in a postmenopausal state. Contraception methods with a reliability exceeding 90 % of common use include cervical caps with spermicide, diaphragms with spermicide, condoms, intra-uterine spirals.
* For the men, are able to conceive - consent to use adequate contraception methods. In the course of the trial, men and their sexual partners should use contraception methods with a reliability exceeding 90 %, or be sterile. Contraception methods with a reliability exceeding 90 % of common use include cervical caps with spermicide, diaphragms with spermicide, condoms, intra-uterine spirals.

Exclusion Criteria:

* A serious post-vaccination reaction (temperature above 40 °C, hyperemia or edema more than 8 cm in diameter) or complications (collapse or shock-like condition that developed within 48 hours after vaccination; convulsions accompanied or not accompanied by a fever due to any previous vaccination);
* Allergic reactions to vaccine components, especially to tetanus toxoid, or to any previous vaccination for the prevention of infections caused by Haemophilus influenza type b;
* Guillain-Barré syndrome (acute polyneuropathy) in the medical history;
* Previous vaccination with rabies vaccines less than 2 months before immunization or scheduled vaccination with rabies vaccines within 1 month after immunization with the trial vaccines;
* Vaccination with any vaccine within one month before the vaccination;
* History of leukemia, tuberculosis, cancer, autoimmune diseases;
* Positive blood test results for HIV, syphilis, hepatitis B/C.
* Volunteers who received immunoglobulin or blood products or had a blood transfusion during the last three months before the trial;
* History of long-term use (more than 14 days) of immunosuppressants or other immunomodulatory products for six months before the trial;
* History of any confirmed or suspected immunosuppressive or immunodeficiency condition;
* History of chronic diseases of the cardiovascular, bronchopulmonary systems, gastrointestinal tract, liver, kidneys, blood in the acute or decompensation stage;
* History of progressive neurological pathology, convulsive syndrome;
* Diabetes, thyrotoxicosis or other diseases of the endocrine system;
* History of eczema;
* Treatment with glucocorticosteroids, including in small doses, as well as local use of products containing steroids;
* According to the medical history, the volunteer was/is a patient of a tuberculosis dispensary and/or narcological dispensary and/or neuropsychiatric dispensary and/or other;
* Acute infectious diseases less than 4 weeks before the start of the trial according to the anamnesis;
* Consumption of more than 10 units of alcohol per week or history of alcohol addiction, product addiction or abuse of pharmaceutical products;
* Smoking of more than 10 cigarettes per day;
* Participation in another clinical trial during the last 3 months;
* Pregnancy or lactation;
* Serious concurrent illnesses or pathological conditions not listed above which, in the opinion of the investigator, could complicate the assessment of the results of the trial including pathological deviations from age norms and laboratory norms of blood and urine parameters, which are clinically significant in the opinion of the investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-06-17 (Actual)

PRIMARY OUTCOMES:
Incidence of local adverse events (AEs) | Days 1-7 post-vaccination
  * Pain at the injection site
  * Hyperemia at the injection site
  * Infiltrate at the injection site
  * Injection site edema
  Severity of an AE was established according to the following classification:
  0 - none - No symptoms
  1. - mild - Mild symptoms
  2. - moderate - Symptoms that disrupt normal daily activities to a certain extent
  3. - severe - Symptoms that disrupt normal daily activities
  Hyperemia/infiltration/edema 0 - none - No symptoms
  1. - mild - Hyperemia with a diameter of up to 50 mm or infiltrate/edema with a diameter of up to 25 mm
  2. - moderate - Hyperemia with a diameter of up to 50 mm or infiltrate/edema with a diameter of 26-50 mm
  3. - severe - Infiltrate/edema more than 50 mm in diameter
Incidence of systemic adverse events (AEs) | Days 1-7 post-vaccination
  Fever, Irritability, Anxiety, Drowsiness, Fainting, Fatigue, Convulsions, Apnea, Arthralgia, Myalgia, Headache, Dizziness, Nausea, Abdominal pain, Loss of appetite, Vomiting, Diarrhea, Rash
  Severity of an AE was established according to the following classification:
  0 - none - No symptoms
  1. - mild - Mild symptoms
  2. - moderate - Symptoms that disrupt normal daily activities to a certain extent
  3. - severe - Symptoms that disrupt normal daily activities
  Fever 0 - none <=37.0°С
  1. - mild > 37.0°С - <=37.5°С
  2. - moderate > 37.6°С - <=38.5°С
  3. - severe > 38.6°С

SECONDARY OUTCOMES:
Incidence of other adverse events (AEs) | Days 8-28 post-vaccination
  0 - none - No symptoms
  1. - mild - Mild symptoms
  2. - moderate - Symptoms that disrupt normal daily activities to a certain extent
  3. - severe - Symptoms that disrupt normal daily activities
Incidence of immediate adverse events (AEs) (allergic reactions) | 2 hours after vaccination
  * Anaphylaxis
  * Quincke's edema
  * Urticaria
    0 - none No symptoms
    1. - mild Mild symptoms
    2. - moderate Symptoms that disrupt normal daily activities to a certain extent
    3. - severe Symptoms that disrupt normal daily activities
Incidence of severe adverse events (SAEs) | Days 0-28
Withdrawal of a volunteer from the trial due to development of an AE/SAE associated with the use of the trial products | Days 0-28
Number of patients with abnormal results of assessment of vital signs - blood pressure (BP) | Days 0-7, 14, 28
  BP measurements include the systolic and diastolic blood pressure, using tonometers
Number of patients with abnormal results of assessment of vital signs - heart rate (HR) | Days 0-7, 14, 28
  HR is measured using a phonendoscope at the apex of the heart (1.5 cm inwards from the left midclavicular line in the 5th intercostal space) during 1 minute.
Number of patients with abnormal results of assessment of vital signs - respiratory rate (RR) | Days 0-7, 14, 28
  RR is counted with a hand placed on the volunteer's chest or abdomen or by holding a stethoscope at the volunteer's nose. The measurement is carried out during one minute.
Number of patients with abnormal results of assessment of vital signs - body temperature | 10 minutes before administration; 20 minutes, 2 hours, 5-8 hours after vaccination; Days 1-7, 14, 28
  Body temperature is measured using a non-contact infrared electronic thermometer.
Number of patients with abnormal results of physical examination | Days 0-7, 14, 28
  Physical examination of volunteers includes an interview, discovery of complaints and symptoms, when required, palpation, auscultation, percussion.
  It is necessary to conduct an examination and (when applicable) palpation, auscultation, percussion for the following organs and systems: skin, mucosa, eyes, oral cavity and pharynx, lungs/chest, heart/cardiovascular system, abdominal organs, nervous system, lymph nodes, musculoskeletal system, thyroid gland. The palpation analysis of lymph nodes (submandibular, cervical, ulnar, inguinal) includes an assessment of their size, consistency, pain, mobility, adhesion between themselves and with surrounding tissues and skin.
Number of patients with abnormal results of neurological status assessment | Days 0,1,3,28
  Assessment of:
  * Cranial nerve function
  * Motor sphere
  * Reflex sphere
  * Sensitive sphere
  * Coordination sphere
  * Pelvic functions
  * Higher mental functions
Number of patients with abnormal ECG findings | Days 0,3
  Standard 12-lead ECG. Assessment of: PQ, QT,QTc intervals, QRS complex
Number of patients with abnormal results of complete blood counts | Days 0,3,14,28
  Red cells, Hemoglobin, ESR, White cells, Differential Leukocyte Count (segmented and rod neutrophils, lymphocytes, monocytes, eosinophils, basophils), Platelets
Number of patients with abnormal results biochemical blood tests | Days 0,3,14,28
  ALT, AST, LDH, Alkaline phosphatase, Bilirubin total, Total protein, Urea, Glucose, C-reactive protein, Creatinine, Prothrombin complex, Cholesterol, В-lipoproteins, Thymol
Number of patients with abnormal results E immunoglobulin tests | Days 0,3,14,28
  Total IgE
Number of patients with abnormal Urinalysis results | Days 0,3,14,28
  pH, Relative density / specific gravity, Protein, Glucose, Red cells, White cells

CONTACTS AND LOCATIONS:
Overall Officials: Ellina Ruzanova, PhD, Study Director — St. Petersburg Research Institute of Vaccines and Sera
Locations (1):
- Federally Funded Healthcare Institution Primary Healthcare Unit No.163, Federal Medical-Biological Agency (FFHI PHU No.163, FMBA of Russia), Коltsovo, Russia